CLINICAL TRIAL: NCT02367326
Title: Identification of Composite Clinical and Lab Scores Associated With a Favorable Clinical Response With Thiopurines in Patients With IBD (Inflammatory Bowel Disease): an International Clinical Trial
Brief Title: Identification of Scores Associated With a Favorable Clinical Response With Thiopurines in IBD Patients
Acronym: SCORE1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Apsen Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1208169; DR-2012-589 (Other: CNIL)
Record Dates: First submitted 2015-02-12; First posted 2015-02-20 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Inflammatory Bowel Diseases
Keywords: score; inflammatory bowel disease; crohn's disease; ulcerative colitis; clinical response; thiopurines
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Inflammatory Bowel Disease: patients with Crohn's Disease or Ulcerative Colitis meeting clinical, endoscopic and histological criteria and on thiopurines at stable doses for at least 3 months, monotherapy or combined with corticotherapy
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection will be carried out by the investigator during a standard hospitalization of the patient

SUMMARY:
Inflammatory bowel disease (IBD) groups together Crohn's Disease (CD) and ulcerative colitis (UC). Its prevalence is high representing approximately 0.4% of the population. The peak incidence for these diseases ranges between 2 and 30 years of age with a second peak for CD recently reported at 60. These diseases develop over time into complications requiring in 2/3 of cases surgical resection procedures in CD and colectomy in over 20% of cases. Cohort data has recently shown that the early use of azathioprine from the first year would decrease the need for surgery. Aside from biologics, azathioprine is the most widely used immunosuppressant in IBD management. Its metabolism is highly variable in the overall population since over 10% of patients are slow metabolizers and 15% fast metabolizers. This explains partly treatment failures and side effects with thiopurines. A lot of research has shown that metabolite measurement of azathioprine (6-TGN end methylated derivatives) could be used clinically even if these results remain controversial. In fact, their positive predicative value (PPV) in clinical response does not exceed 60%. This costly testing cannot be done everywhere, is not reimbursed by national health services, and may not be used in some countries. It is, however, key in order optimize these drugs at a time when only two anti-TNFs are possible in the event of failure on thiopurines. Older studies have shown that MCV and lymphonenia could be markers for thiopurine impregnation. Recently, an American study provided a mathematic formula enabling to achieve over 80% PPV for the clinical response on AZA but this calculation needs to be confirmed and it is, moreover, patented (costly).

DETAILED DESCRIPTION:
We suggest developing a predictive score for clinical thiopurines in IBD based on routine lab data obtained when monitoring patients on thiopurines. This initial work will enable to identify clinical and/or lab factors in order to develop a score based on an international, multicenter, cross-section study. Two hundred patients with treatment failure on thiopurines will be included and at least as many in clinical remission on thiopurines. A subsequent longitudinal study, over all recruiting centers will enable to validate the score. Finally, a prospective study will assess the clinical impact of the optimization of this score in patients sustaining a treatment failure on thiopurines. This score - if confirmed - will subsequently be at no additional cost in the management of patients on thiopurines.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients affiliated with or beneficiaries of a national health insurance scheme
* Male our female over 18 years of age and under 70 having given his/her informed consent to participate in this trial.
* Any patients with Crohn's Disease or Ulcerative Colitis meeting clinical, endoscopic and histological criteria.
* Patients on thiopurines at stable doses for at least 3 months, monotherapy or combined with corticotherapy using the following doses:

AZATHIOPRINE at the dose of 2 to 2.5 mg/kg/day, regular oral dosing for 3 months or PURINETHOL at the dose of 1 to 1.5 mg/kg/day, regular oral dosing for 3 months

Exclusion Criteria:

* Patients with intolerance to thiopurines resulting in reduction or discontinuation of thiopurines by the referring physician.
* Post operative Crohn's Disease patients for whom thiopurines were indicated preventively or in the event of endoscopic abnormalities.
* Extensive colic resection, (sub)total colectomy.
* History of > 3 resections of the small intestine or diagnosis of a short bowel
* Crohn's Disease with a perianal lesion whether the latter is isolated or the focus of the disease
* Patient with a enterocutaneous, abdominal or pelvic fistula with abscess or fistula likely to require surgery during the study
* Ileostomy, colostomy or known intestinal stenosis
* Severe active infection
* Active neoplasia
* Known TPMPT homozygote mutation
* Patients on anti-TNF or Methotrexate in the last 3 months or during thiopurine therapy
* Patients on Allopurinol.
* Patient who expressed his/her refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Crohn's Disease or Ulcerative Colitis and on thiopurines at stable doses for at least 3 months, monotherapy or combined with corticotherapy
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
number of patient with therapeutic failure on thiopurines | day 0 (inclusion)
  A therapeutic failure on thiopurines will be considered to be any patient with at least one of the following criteria:
  * For Crohn's Disease: a HBI score > 4
  * For Ulcerative Colitis: a partial Mayo score > 2 or activity reported by the expert at the time of a visit
  * For both disease:
    * Corticodependence, defined according to ECCO criteria, as an impossibility to reduce the dose of Prednisolone to less than 10 mg/day (or 3 mg/day for Budesonide) in the 3 months following corticotherapy induction.
    * Corticoresistance, defined according to ECCO criteria, as a lack of response to the dose of 0.75mg/kg of a Prednisone equivalent for 4 weeks.
    * the need to change treatment or a surgical indication.

SECONDARY OUTCOMES:
number of patient in clinical remission on thiopurines | day 0 (inclusion)
  A clinical remission shall be considered as any patients with at least one of the following criteria:
  * For Crohn's Disease: a HBI score < 4
  * For ulcerative colitis: a partial Mayo score ≤ 2 with no subscore > 1
  * For both diseases, no corticotherapy for at least 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier ROBLIN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (15):
- France (15):
  - CHU Jean Minjoz, Besançon
  - CHU Caen, Caen
  - CHU Dijon, Dijon
  - CHRU Lilles, Lilles
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes - Hôtel-Dieu, Nantes
  - CHU Nice, Nice
  - CHR Orléans, Orléans
  - Hôpital Saint-Antoine, Paris
  - CHU Bordeaux, Pessac
  - CH Lyon Sud, Pierre-Bénite
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Saint-Etienne, Saint-Etienne